CLINICAL TRIAL: NCT05421221
Title: A Randomized Controlled Trial of the Effectiveness of Olfactory Training on Loss of Smell Related to COVID-19 (SMELL)
Brief Title: Olfactory Training in COVID-19 Associated Loss of Smell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12732020
Record Dates: First submitted 2022-06-15; First posted 2022-06-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Hyposmia
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olfactory training group (Experimental): 12 weeks of olfactory traiing with Sniffin' sticks "Duftquartett".
  Interventions: Device: Sniffin' sticks Duftquartett
- no olfactory training with natural history of the disease (No Intervention): natural history of the disease

INTERVENTIONS:
Device: Sniffin' sticks Duftquartett — 4-odor training set over 12 weeks with Sniffin' sticks "Duftquartett"
  Arms: olfactory training group

SUMMARY:
Olfactory dysfunction (OD) like hyposmia or anosmia has been realized as a common symptom or even cardinal sign of the disease and can be persisting after recovering.

There are two different hypotheses on the pathogenesis of OD in past COVID-19: The central hypothesis, which speculates on neurotrophic abilities on olfactory receptors in the neuroepithelium, and the peripheral hypothesis, which speculates on damage of the sensory olfactory epithelium.

Potential treatment strategies aim for the unique neural plasticity of the olfactory system and its potential for recovery.

Clinical studies and case reports have shown a promising effect of olfactory training (OT) by frequent sniffing and/or exposure to odors 2-4 times a day for several weeks.

The main objective of the study is to assess the effects of olfactory training in patients with COVID-19 related OD on:

1. objective olfactory testing with the Sniffin' sticks test (identification and discrimination),
2. subjective OD and its impact on the daily life,
3. other clinical scales and questionnaires referring to OD-related mood and quality of life,
4. gender differences in COVID-19 related OD. Approach / methods OT will be performed twice a day with a 4-odor training set for 12 weeks. Effects of OT on COVID-19 related OD will be measured with objective and subjective efficacy variables.

The sense of smell is an important function for social relationships and is therefore a challenging clinical problem with few proven therapeutic options.

With this new approach, we want to investigate a possible simple treatment for an impedimental symptom of COVID-19, but also learn more about the pathomechanism of post-infectious OD.

To our knowledge, this will be the first study comparing patients with COVID-19 associated OD with and without OT in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged over 18 years;
* confirmed diagnosis of COVID-19 at least three months ago (history of positive PCR-testing required) or positive serum nucleocapsid antibody titer against SARS-CoV2;
* post-infectious COVID-19 related olfactory dysfunction persisting for at least three months with abnormal Sniffin' sticks test (<13/16 items correct in the identification part);
* the patient is willing to undergo odor training over 12 weeks;
* written ICF is obtained.

Exclusion Criteria:

* History of olfactory dysfunction prior to COVID-19 infection due to other conditions e.g. status post traumatic brain injury, Parkinson's disease, allergic rhinitis, etc.;
* Nasal pathology not related to COVID-19 in the systematic otorhinolaryngological examination including endoscopy.
* the participant is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
primary endpoint | 12 weeks
  changes between groups from baseline to week 12/termination visit regarding correct odor identification and discrimination

SECONDARY OUTCOMES:
Visual Analog Scale | 12 weeks
  from 0 to 10, higher score means better subjective olfaction
Short-Form-36 Health Survey Questionnaire (SF-36) | 12 weeks
  Quality of Life Each domain is scored from 0 to 100, higher scores mean better health status
Mood inventory | 12 weeks
  Will be applied in German
Hospital Anxiety and Depression Scale | 12 weeks
  Anxiety and Depression Each item is scored on a 4-point scale from 0 to 3; lower scores mean less anxiety/depression
Patient Progress and treatment response over time | 12 weeks
  Using Patient Global Impression of Improvement
Clinical treatment response over time | 12 weeks
  Using Clinical Global Impression of Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Heim, MD PhD, Study Chair — Medical University of Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Yes
Data supporting the results will be archived in an appropriate public repository
Supporting Information: Study Protocol
Time Frame: after publication of the primary data
Access Criteria: data will be deposited in appropriate public repositories

REFERENCES:
- [Derived] De Cleene N, Jagusch F, Schmutzhard J, Gottfried T, Peball M, Djamshidian A, Ellmerer P, Goebel G, Helbok R, Kindl P, Loffler-Ragg J, Weiss G, Seppi K, Heim B; SMELL study-group. Protocol for olfactory training in persisting COVID-19-associated loss of smell (SMELL): a monocentric randomised controlled trial conducted in Innsbruck. BMJ Open. 2025 May 27;15(5):e094027. doi: 10.1136/bmjopen-2024-094027. PMID 40436445